CLINICAL TRIAL: NCT06081764
Title: Investigation of the Effects of Physical Activity on Physical Fitness Parameters, Functional Fitness Age and Quality of Life in Women at Risk of Osteoporosis
Brief Title: Investigation of the Effects of Physical Activity in Women at Risk of Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatma Nur Alçın, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03.12.2021-E.136626
Record Dates: First submitted 2023-08-25; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis Risk
Keywords: Functional Fitness Age; Osteoporosis; Otago Exercise Program; Post-Menopausal Woman; Quality of Life; Physical Fitness
MeSH Terms: conditions — Osteoporosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): They participated the Otago Exercise Program, which last 3 days a week and an average of 30 minutes per day for 12 weeks in total. In addition, they did moderate-intensity walking exercise for 30 minutes a day, 2 days a week.
  Interventions: Other: Exercise
- Control Group (No Intervention): No program were applied to the participants in the control group.

INTERVENTIONS:
Other: Exercise — Doing Otago Exercise Program, which lasting 3 days a week and an average of 30 minutes per day under the supervision of a physiotherapist. Also doing walking exercise for 30 minutes a day, 2 days a week for total of 12 weeks.
  Arms: Otago Exercise Program

SUMMARY:
The goal of this clinical trial is to investigate the effects of the increase in the physical activity level of women at risk for osteoporosis in the post-menopausal period on the physical fitness, functional fitness age and quality of life. The main question it aims to answer is:

• Does the increase in the level of physical activity positively affect the physical fitness parameters (strength, endurance, balance, agility and flexibility), functional fitness ages and quality of life of post-menopausal women with moderate to high osteoporosis risk?

Participants in the intervention group were given the Otago Exercise Program, which will last 3 days a week and an average of 30 minutes per day for 12 weeks. The exercises were done one-by-one with a physiotherapist. No program were applied to the participants in the control group, and they were asked to continue their daily living activities in the same way.

Researchers will compare two groups to see if there is a difference in effects of Otogo Exercise Program on physical fitness, functional fitness age, and quality of life.

DETAILED DESCRIPTION:
The osteoporosis risks of the participants were calculated according to the Osteoporosis Self-Assessment Tool for Women (OST). Women have medium and high risk were included in the study.

Otago Exercise Program includes strengthening exercises consisting of knee extension, knee flexion, hip abduction, ankle dorsi flexion, and 12 balance exercises consisting of plantar flexion and squatting, walking backward, walking and rolling back, sideways walking, tandem stance, tandem gait, standing on one leg, heels walking on toes, walking on tiptoe, sitting and standing, climbing and descending stairs, and backward tandem walking.

• In addition, moderate-intensity walking exercise for 30 minutes a day, 2 days a week, was recommended to the patients in experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Being at medium-high risk as a result of the Osteoporosis Self-Assessment Tool for Women (OST)
* Being 54 years old and over
* Being in the post-menopausal period

Exclusion Criteria:

* Having a broken history
* Having a history of surgery in the last 1 year
* Having a cognitive or physical condition that will prevent them from exercising
* Exercising regularly for more than 30 minutes a day, at least 3 days a week

Ages: 54 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female individuals were included in the clinical trial.
Enrollment: 40 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Strength | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Lower extremity strength will be evaluated with the 30-second sit-stand test included in the ''Senior Fitness Test'', which is a physical fitness assessment tool.
Upper Extremity Strength | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Upper extremity strength will be evaluated with the 30-second elbow bend test included in the ''Senior Fitness Test'', which is a physical fitness evaluation tool.
Aerobic Endurance | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Aerobic endurance will be evaluated with the 2-minute walking test included in the ''Senior Fitness Test'', which is a physical fitness evaluation tool.
Upper Extremity Flexibility | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Upper extremity flexibility will be evaluated with the sit-reach test and back scratching test included in the ''Senior Fitness Test'', which is a physical fitness evaluation tool.
Agility | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Agility will be evaluated with the stand-up and walk test included in the ''Senior Fitness Test'', which is a physical fitness evaluation tool.
Quality of Life of Individual | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  Quality of Life was tested with the ''Quality of Life for Osteoporosis Questionnaire''. The scale consists of 41 questions. There are 5 subscales: pain (5 items), physical function (17 items), social activity (7 items), general health assessment (3 items) and mental function (9 items). For each subgroup and total result in the scale, 0 points indicate the best health status, while higher scores indicate poor quality of life.

SECONDARY OUTCOMES:
Dynamic Balance | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  In addition to evaluating agility with the standing and walking test included in the "Senior Fitness Test", which is a physical condition evaluation tool, dynamic balance will also be evaluated since this test is an indicator of dynamic balance.

OTHER OUTCOMES:
Physical Activity Level | The first measurement was made just before the start of the treatment, and the second measurement was made just after the end of the treatment.
  The physical activity levels of the participants were evaluated with the Global Physical Activity Questionnaire. This survey, consisting of a total of 16 questions, evaluates physical activity participation in 3 different areas. These areas; work-related, transfers (walking, cycling) and leisure activities. Calculation of the total score includes the sum of the duration (minutes) and frequency (days) of walking, moderate activity and vigorous activity. The energy required for activities is calculated with the MET-minute score. An increase in this score indicates that the daily and weekly physical activity level increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Çetişli Korkmaz, Prof., Study Director — Pamukkale University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Gölhisar, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wen HJ, Huang TH, Li TL, Chong PN, Ang BS. Effects of short-term step aerobics exercise on bone metabolism and functional fitness in postmenopausal women with low bone mass. Osteoporos Int. 2017 Feb;28(2):539-547. doi: 10.1007/s00198-016-3759-4. Epub 2016 Sep 9. PMID 27613719
- [Background] Latorre-Rojas EJ, Prat-Subirana JA, Peirau-Teres X, Mas-Alos S, Beltran-Garrido JV, Planas-Anzano A. Determination of functional fitness age in women aged 50 and older. J Sport Health Sci. 2019 May;8(3):267-272. doi: 10.1016/j.jshs.2017.01.010. Epub 2017 Jan 23. PMID 31193284
- [Background] Subramaniam S, Ima-Nirwana S, Chin KY. Performance of Osteoporosis Self-Assessment Tool (OST) in Predicting Osteoporosis-A Review. Int J Environ Res Public Health. 2018 Jul 9;15(7):1445. doi: 10.3390/ijerph15071445. PMID 29987247
- [Background] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194